CLINICAL TRIAL: NCT03680209
Title: Interest of Training in Procedural Simulation of Nurses in Reducing Complications Related to Arteriovenous Fistula Puncture in Chronic Hemodialysis Patients
Brief Title: Training Procedural Simulation of Nurses in Reducing Complications Related to Arteriovenous Fistula Puncture
Acronym: SIMFAV
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A00072-53
Record Dates: First submitted 2018-06-13; First posted 2018-09-21 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2018-09

CONDITIONS: Nurse's Role; Simulation; Arteriovenous Fistula
Keywords: Task trainning; Procedural simulation
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Simulation — pre-training observation training post training observation

SUMMARY:
Interest of training in procedural simulation of nurses in the reduction of complications related to arteriovenous fistula puncture in hemodialysis patients

DETAILED DESCRIPTION:
Primary objective :

To compare the number of complications related to arteriovenous fistula (AVF)puncture before and after a complete simulation training program, on a fistula arm of procedural simulation (conceptualization of the approach + puncture + palpation + identification + use of ultrasound)

Secondary objective (s):

Compare other adverse events related to AVF puncture during a hemodialysis session

ELIGIBILITY:
Inclusion Criteria:

* Patients whose nurse is trained in hemodialysis receiving a FAV puncture in the hemodialysis unit of the nephrology department, dialysis, transplantation

Exclusion Criteria:

* Patients with AVF puncture in the emergency / withdrawal area of the nephrology department, dialysis, transplantation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients who come to dialysis
Sampling Method: Non-Probability Sample
Enrollment: 1280 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Complications related to arteriovenous fistula puncture (AVF) | 25 days
  Number of complications of fistula puncture :
  either failed unipuncture puncture either failed bipunctional puncture either simple hematoma either hematoma does not allow the continuation of dialysis

SECONDARY OUTCOMES:
Adverse events related to AVF puncture during a hemodialysis session | 25 days
  Number of perdialytic bleeding : accidental removal of the needle
Adverse events related to AVF puncture during a hemodialysis session | 25 days
  Pain score (EN digital scale) felt at the time of puncture

CONTACTS AND LOCATIONS:
Overall Officials: Erwan Guillouët, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided
Publication